CLINICAL TRIAL: NCT01112098
Title: Randomized Trial of a Mailed Intervention and Self-Scheduling to Improve Osteoporosis Screening in Postmenopausal Women
Brief Title: Improving Quality of Osteoporosis Care Through Patient Storytelling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Jeffrey R. Curtis, MD MPH, UAB
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: X070502003
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Educational Pamphlet and letter (Experimental): Letter invites patient to self-schedule a DXA; educational pamphlet includes information about DXA scans
  Interventions: Behavioral: Patient Pamphlet

INTERVENTIONS:
Behavioral: Patient Pamphlet — letter informs patient of opportunity to self-schedule a DXA scan; pamphlet includes information about receiving a DXA scan
  Other Names: Educational Materials; Written Materials; Mailed Letter

SUMMARY:
The purpose of this exploratory study is to test novel, mailed, low-cost, direct-to-patient intervention materials (i.e., a personalized letter and osteoporosis information pamphlet) designed to increase rates of dual energy X-ray absorptiometry (DXA) utilization and improve osteoporosis quality of care.

DETAILED DESCRIPTION:
While the occurrence of a fragility fracture (e.g. hip fracture) is indicative of low BMD and a clinical diagnosis of osteoporosis made, osteoporosis can be identified in asymptomatic patients using dual energy x-ray absorptiometry (DXA). United States (U.S.) guidelines recommend screening bone density tests using central DXA in all women 65 years or older. However, fewer than one-third of eligible U.S. women age 65 and older undergo DXA testing. The main barrier to achieving greater rates of osteoporosis screening is identifying a systematic, effective, and generalizable way for healthcare providers and patients to schedule DXA results.

Given that national guidelines recommend DXA screening for all older women, the reasons a majority of women do not receive DXA testing are likely multifactorial. Patients and their health care providers may be unaware of preventative screening recommendations and the reasons for these recommendations. Screening tests that are required relatively infrequently (i.e. less than once a year) may be difficult for patients and physicians to remember if there are few triggers (e.g. seasonality as a trigger to motivate influenza vaccination). Additionally, primary care providers (PCPs) are responsible for managing a large number of comorbidities and acute care needs and may be unable to stay current with all preventative care needs during increasingly short clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 65 or older
* At least one visit with a primary care physician in the previous 12 months

Exclusion Criteria:

* DXA scan in the previous 5 years

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2997 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
DXA scheduled | 6 months
  Patient scheduled a DXA within 6 months of receiving intervention materials

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Curtis, MD, MPH, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Warriner AH, Outman RC, Kitchin E, Chen L, Morgan S, Saag KG, Curtis JR. A randomized trial of a mailed intervention and self-scheduling to improve osteoporosis screening in postmenopausal women. J Bone Miner Res. 2012 Dec;27(12):2603-10. doi: 10.1002/jbmr.1720. PMID 22836812